CLINICAL TRIAL: NCT01348607
Title: A Randomized, Phase II Placebo-controlled Study of the Use of Extended-release Methylphenidate or Modafinil for the Treatment of Excessive Daytime Sleepiness in Children Following Cancer Therapy
Brief Title: Methylphenidate HCl or Modafinil in Treating Young Patients With Excessive Daytime Sleepiness After Cancer Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study only randomized 1 subject and was determined not feasible by DSMB
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SCUSF 0803; SCUSF-0803 (Other: SunCoast CCOP Research Base); 5U10CA081920-11 (NIH)
Record Dates: First submitted 2011-05-04; First posted 2011-05-05 (Estimated); Results first posted 2013-09-19 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-01

CONDITIONS: Central Nervous System Tumor, Pediatric; Fatigue; Specific Disorders of Sleep
Keywords: psychosocial effects of cancer and its treatment; sleep disorders; fatigue; childhood craniopharyngioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Fatigue; Sleep Wake Disorders | interventions — Methylphenidate; Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I - methylphenidate hydrochloride (Experimental): Patients receive oral methylphenidate extended-release once daily for 7-42 days in the absence of unacceptable toxicity.
  Interventions: Drug: methylphenidate hydrochloride
- Arm II -modafinil (Experimental): Patients receive oral modafinil once daily for 7-42 days in the absence of unacceptable toxicity.
  Interventions: Drug: modafinil
- Arm III placebo (Placebo Comparator): Patients receive oral placebo once daily for 7-42 days in the absence of unacceptable toxicity.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: methylphenidate hydrochloride — Given orally
  Other Names: methylphenidate HCl; Concerta
  Arms: Arm I - methylphenidate hydrochloride
Drug: modafinil — Given orally
  Other Names: Provigil
  Arms: Arm II -modafinil
Drug: placebo — Given orally
  Other Names: potato starch placebo; placebo capsule
  Arms: Arm III placebo

SUMMARY:
RATIONALE: Methylphenidate hydrochloride or modafinil may help reduce daytime sleepiness and improve the quality of life of patients with excessive daytime sleepiness after cancer therapy. It is not yet known whether methylphenidate hydrochloride or modafinil are more effective than a placebo in reducing daytime sleepiness in these patients.

PURPOSE: This randomized phase II trial is studying methylphenidate hydrochloride or modafinil to see how well they work compared with a placebo in treating young patients with excessive daytime sleepiness after cancer therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of methylphenidate hydrochloride and modafinil to placebo in pediatric patients with excessive daytime sleepiness following cancer therapy.

Secondary

* Compare the efficacy of half dose methylphenidate hydrochloride and modafinil to placebo in these patients.
* Assess the effects of these regimens on daytime sleepiness as measured by the Pediatric Daytime Sleepiness Scale or the Cleveland Adolescent Sleepiness Questionnaire.
* Assess the effects of somnolence symptoms on fatigue as measured by the PedsQL Multidimensional Fatigue Scale.
* Assess the effects of somnolence symptoms on the quality of life as measured by the PedsQL Quality of Life Inventory 4.0.
* Determine the incidence of side effects associated with these regimens.
* Determine the prevalence of sleep complaints as measured by the Pediatric Sleep Questionnaire. (Exploratory)

OUTLINE: This is a multicenter study. Patients are stratified according to age (8-10 years vs 11-12 years vs 13-17 years vs 18-25 years). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive oral methylphenidate hydrochloride extended-release once daily for 7-42 days in the absence of unacceptable toxicity.
* Arm II: Patients receive oral modafinil once daily for 7-42 days in the absence of unacceptable toxicity.
* Arm III: Patients receive oral placebo once daily for 7-42 days in the absence of unacceptable toxicity.

Patients or their parents complete age-specific sleep and quality-of-life questionnaires at baseline and after completion of treatment. Patients or their parents complete daily sleep diaries during the study to collect information about the date, type of day (school, weekend, or vacation), hours of sleep, anytime the actigraph was removed during the day, time the child went to bed, and time the child got out of bed in the morning. Patients are also instructed to wear an actigraph on their non-dominant wrist for 1 week before starting treatment and during the first and last week of treatment (3 weeks total) to assess sleep-wake patterns.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patient and family must agree to return to the clinic up to 8 times within 2 months
* Children ≥ 8 and <18 years of age at the time of study entry who were previously treated for:
* a hypothalamic tumor
* mid-line brain tumor
* a tumor involving one or both thalami
* craniopharyngioma
* diagnosis of hydrocephalus secondary to a brain tumor or treatment of a brain tumor that required placement of a permanent shunt.
* Off cancer treatment for at least six months
* Proficient in English
* Able to swallow capsules
* Experiencing symptoms of excessive daytime sleepiness (EDS) for at least three months prior to study entry that is not a result of inadequate sleep hygiene or other known medical disorder.
* Negative pregnancy test

EXCLUSION CRITERIA:

* Patients treated with doxorubicin or high dose cyclophosphamide
* History of a clinically significant drug sensitivity to methylphenidate, modafinil, armodafinil or any of their components
* Known cardiac disorders including arrhythmias, hypertension requiring treatment or structural heart disease
* Have taken methylphenidate or modafinil within the last 14 days
* Current/concurrent use of antihistamines, benzodiazepine, anticonvulsants or alcohol
* Clinical diagnosis of major depression, subclinical depression, or anxiety disorder
* History of psychosis or mania
* Patients with suicidal ideation
* Diagnosis with anemia, untreated hypothyroidism, mononucleosis or narcolepsy
* History of substance abuse
* Pregnant or breast feeding
* A total dietary intake of more than 500 mg of caffeine per day (e.g., approximately ten 330 mL cans of soft drinks, five cups of coffee or tea, or 750 g chocolate per day).

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2010-07; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Rosen, MD, Study Chair — Children's Hospitals and Clinics of Minnesota - St. Paul; Tom Geller, MD, Study Chair — St. Louis University

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I - Methylphenidate Hydrochloride | Arm II -Modafinil | Arm III Placebo
Started | 1 | 0 | 0
Completed | 1 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I - Methylphenidate Hydrochloride | Arm II -Modafinil | Arm III Placebo | Total
Number analyzed (Participants) | 1 | 0 | 0 | 1
Age, Categorical [Number; unit: participants]
  <=18 years | 1 |  |  | 1
  Between 18 and 65 years | 0 |  |  | 0
  >=65 years | 0 |  |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.9 |  |  | 13.9
Gender [Number; unit: participants]
  Female | 0 |  |  | 0
  Male | 1 |  |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Average Daytime Napping Minutes in a Week
Description: Outcome measure was the total of daytime napping minutes in a week as assessed by participant sleep diaries
Time Frame: 29 days
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Arm I - Methylphenidate Hydrochloride | Arm II -Modafinil | Arm III Placebo
Number analyzed (Participants) | 1 | 0 | 0
minutes | 36.7 |  |

2. Secondary Outcome: Adverse Events
Description: Adverse events assessed at all subject visits by interviews with the subject and the subject's parent/ primary caregiver.
Time Frame: 29 days
Measure: Number; unit: events
Arm/Group | Arm I - Methylphenidate Hydrochloride | Arm II -Modafinil | Arm III Placebo
Number analyzed (Participants) | 1 | 0 | 0
events | 1 |  |

ADVERSE EVENTS:
Time Frame: 1 month
Description: Complete and frequent monitoring for adverse events (AEs) were incorporated using the Systematic Assessment for Treatment Emergent Effects (SAFTEE),developed by the National Institute of Mental Health. AEs will also be assessed by weekly physical exam, review of patient/caregiver daily sleep and medicine logs and patient/caregiver interview.
Arm/Group | Arm I - Methylphenidate Hydrochloride | Arm II -Modafinil | Arm III Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Methylphenidate Hydrochloride (N=1) | Arm II -Modafinil (N=0) | Arm III Placebo (N=0)
decreased appetite (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was closed prior to completion due to a lack of feasibility and low accrual by the Data Monitoring and Safety Board (DSMB).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No